CLINICAL TRIAL: NCT03029481
Title: Single Patient Expanded Access to Ganitumab for Metastatic Ewing Sarcoma
Status: No longer available | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-000019; JCCCID738 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — ganitumab

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Ganitumab — The patient will receive ganitumab, 18 mg/kg/dose intravenously every 2 weeks until clinical progression or decision to move to an alternate therapy.
  Other Names: AMG 479

SUMMARY:
Despite improvements in outcomes for patients with localized Ewing sarcoma, patients with relapsed metastatic Ewing sarcoma continue to have poor outcomes with current chemotherapy options. A large body of preclinical data supports a role for IGF-1R inhibition in the treatment of Ewing sarcoma.

More recently, clinical trials of IGF-1R monoclonal antibodies have demonstrated single- agent activity in patients with relapsed Ewing sarcoma. Ganitumab (AMG 479) is a fully human monoclonal antibody directed against IGF-1R. We are proposing this single-agent expanded access IND to provide our patient the opportunity to benefit from this treatment after having developed progressive disease after multiple lines of prior therapy.

DETAILED DESCRIPTION:
Despite improvements in outcomes for patients with localized Ewing sarcoma, patients with relapsed metastatic Ewing sarcoma continue to have poor outcomes with current chemotherapy options. A large body of preclinical data supports a role for IGF-1R inhibition in the treatment of Ewing sarcoma.

More recently, clinical trials of IGF-1R monoclonal antibodies have demonstrated single- agent activity in patients with relapsed Ewing sarcoma. Ganitumab (AMG 479) is a fully human monoclonal antibody directed against IGF-1R. We are proposing this single-agent expanded access IND to provide our patient the opportunity to benefit from this treatment after having developed progressive disease after multiple lines of prior therapy.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: Confirmed translocation-positive Ewing sarcoma

Organ Function Requirements:

Serum creatinine < 1.4 Adequate liver function

* Total bilitubin <1.5x upper limit of normal for age
* SGPT (ALT) < 5x upper limit of normal for age Adequate cardiac function > 50% by echocardiogram Bone Marrow
* Absolute neutrophil count > 750
* Platelet count > 75

Exclusion Criteria:

* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained. Lactating females are not eligible unless they have agreed not to breastfeed their infants for the duration of protocol therapy. Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of protocol therapy.
* Patients with known pre-existing diabetes mellitus will be excluded from study.

Ages: 48 Years to 50 Years | Sex: All
Age Groups: Adult